CLINICAL TRIAL: NCT01975571
Title: Iowa Cochlear Implant Clinical Research Center Hybrid Cochlear Implants in Severe to Profound Adults, Children, and Adolescents
Brief Title: Hybrid Cochlear Implants in Severe to Profound Adults, Children, and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce J Gantz (Other)
Responsible Party: Sponsor-Investigator, Bruce J Gantz, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201106758
Record Dates: First submitted 2012-07-06; First posted 2013-11-04 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Hearing Loss, High-Frequency
Keywords: residual hearing; hybrid; hearing preservation
MeSH Terms: conditions — Hearing Loss, High-Frequency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adult (Experimental): Population 1: 15 Adults who have a severe sensorineural hearing loss with a pure-tone average (PTA) between 60-90 dB HL between 125-1500 Hz and profound loss at higher frequencies.
  Intervention: These patients will receive a Hybrid L24 cochlear implant.
  Interventions: Device: Cochlear® Nucleus™ Hybrid L24
- Children and adolescents (L24) (Experimental): Children (ages 5-12 years) and adolescents (ages 13-15 years) who have a sensorineural hearing loss with a pure-tone average (PTA) between 70-90 dB HL between 125-1500 Hz, a hearing threshold >90 dB HL at 1500 Hz and profound loss at higher frequencies.
  Intervention: These patients will receive a Hybrid L24 cochlear implant.
  Interventions: Device: Cochlear® Nucleus™ Hybrid L24
- Children and adolescents S12 (Experimental): Children (ages 5-12 years) and adolescents (ages 13-15 years) who have a sensorineural hearing loss with a pure-tone average (PTA) between 70-90 dB HL between 125-1500 Hz, a hearing threshold hearing threshold between 70-90 dB HL at 1500 Hz and profound loss at higher frequencies.
  Intervention: These patients will receive a Hybrid S12 cochlear implant.
  Interventions: Device: Cochlear® Nucleus™ Hybrid S12

INTERVENTIONS:
Device: Cochlear® Nucleus™ Hybrid L24 — The Nucleus Hybrid L24 cochlear implant incorporates an electrode array designed to preserve residual hearing. This has been accomplished by employing a thin, straight, intracochlear electrode array attached to a Nucleus cochlear implant receiver/stimulator. The Nucleus Hybrid L24 array has 22 electrodes spread over 16 mm and an anticipated insertion depth of 16 mm. It is slim, with its dimensions ranging from 0.35 x 0.25 mm (at the tip) to 0.55 x 0.4 mm, and designed to minimize lateral wall forces with a stiffened basal section to prevent buckling. The resultant insertion angle is about 280-300° in the scala tympani for the Hybrid L24, as confirmed in temporal bone trials at the Medical University Hannover and the University of Melbourne.
  Arms: Adult; Children and adolescents (L24)
Device: Cochlear® Nucleus™ Hybrid S12 — The Nucleus Hybrid S12 cochlear implant incorporates an electrode array designed to stimulate the high-frequency, basal region of the cochlea while maintaining useful acoustic hearing in the low-frequency, apical region. This has been accomplished by employing a short, thin, straight intracochlear electrode array attached to a Nucleus cochlear implant receiver/stimulator. The electrode array incorporates a collar to prevent over-insertion, or further migration, into the cochlea beyond the point where the basal turn curves into the ascending segment. Thus, the electrode array is placed within the straight segment of the basal turn of the scala tympani via a cochleostomy.
  Arms: Children and adolescents S12

SUMMARY:
The purpose of this study is to determine if adults and children with residual low-pitch hearing in the severe hearing loss range can develop improved speech perception by combining their residual acoustic hearing with electrical stimulation through a short cochlear implant. The low-pitches would be amplified with a hearing aid and the high-pitch sounds would be stimulated electrically.

DETAILED DESCRIPTION:
The purpose of this study is to determine if individuals with residual low-frequency hearing in the severe range can develop improved speech perception by combining their residual acoustic hearing with electrical processing through a cochlear implant designed to stimulate the high-frequency basal and middle turn of the cochlea while preserving useful low-frequency acoustic hearing. To accomplish this, we propose to implant individuals with severe hearing with a Cochlear® Nucleus™ Hybrid L24 Implant or a Cochlear® Nucleus™ Hybrid S12 in the poorer ear. We believe these devices will do less damage to the Organ of Corti structures, than longer, more invasive standard cochlear implant electrodes.

Two different populations will be studied under this IDE.

Population 1: 15 Adults who have a severe sensorineural hearing loss with a pure-tone average (PTA) between 60-90 decibels (dB) hearing level (HL) between 125-1500 Hz and profound loss at higher frequencies will be implanted with the Cochlear® Nucleus™ Hybrid L24 Implant. The potential subject will present with Consonant-Nucleus-Consonant (CNC) monosyllabic word scores between 0-35% in the ear to be implanted and up to 60% understanding in the contralateral ear in the best-aided condition.

Population 2: 30 Children (ages 5-12 years) and adolescents (ages 13-15 years) who have a sensorineural hearing loss with a pure-tone average (PTA) between 60-90 dB HL between 125-1500 Hz and profound loss at higher frequencies will be implanted with the Cochlear® Nucleus™ Hybrid L24 Implant or the Cochlear® Nucleus™ Hybrid S12 Implant. Those that have hearing thresholds between 60-90 dB HL at 1500 Hz would be implanted with the less invasive shorter 10 mm Hybrid S12 in attempt to better preserve the middle frequency range. Those with hearing thresholds >90 dB HL at 1500 Hz would receive the longer 16 mm Hybrid L24 electrode. The potential subject will present with Phonetically Balanced Kindergarten (PB-K) monosyllabic word scores between 0-50% in the ear to be implanted and up to 60% understanding in the contralateral ear in the best-aided condition.

Through the preserved acoustic hearing, we believe the subject will experience better signal to noise ratios for speech perception in noise, better localization of sound and an improvement music perception. Histological evidence from patients implanted with standard arrays and our experience with a short electrode array for implantation of individuals with significant residual hearing both support this assumption (Nadol, Shiao, Burgess, Ketten, Eddington et al., 2001). The duration of this study will be 2 years (24 months) for adults and for 5 years (60 months) in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

1.1 Criteria for Inclusion in Population 1

Criterion for selection will be subject interest in preservation of residual hearing; severe sensorineural hearing loss; lack of benefit from appropriately fit binaural hearing aids worn on a full-time basis; and realistic expectations. Qualified participants must also meet the following criteria for inclusion:

1. Eighteen year of age or older at the time of implantation.
2. Severe sensorineural hearing loss with a pure-tone average (PTA) between 60-90 dB HL between 125-1500 Hz and profound loss at higher frequencies in the ear to be implanted.
3. Speech Perception:

   * The Consonant-Nucleus-Consonant (CNC) word recognition score between 0% and 35% inclusive in the ear to be implanted.
   * The CNC word recognition score in the contralateral ear equal to or better than, in the ear to be implanted but not more than 60% in the best-aided condition.
4. English spoken as a primary language.
5. Willingness to comply with all study requirements.
6. Minimum of 30 day hearing aid trial with appropriately fit hearing aids worn on a full-time basis (8 hours per day).
7. Patent cochlea and normal cochlear anatomy.

1.2 Criteria for Inclusion in Population 2

Criterion for selection will be parent interest in preservation of residual hearing; severe post-lingual onset of sensorineural hearing loss; lack of benefit from appropriately fit binaural hearing aids worn on a full-time basis; and supportive family dynamics. Qualified participants must also meet the following criteria for inclusion:

1. Five to fifteen years of age at the time of implantation.
2. Severe sensorineural hearing loss with a pure-tone average (PTA) between 60-90 dB HL between 125-1500 Hz and profound loss at higher frequencies in the ear to be implanted.
3. Speech Perception:

   * The Phonetically Balanced-Kindergarten (PB-K) word recognition score between 0% and 50% inclusive in the ear to be implanted.
   * The PB-K word recognition score in the contralateral ear equal to or better than, in the ear to be implanted but not more than 60%.
4. English spoken as a primary language.
5. Willingness to comply with all study requirements.
6. Minimum of 30-day hearing aid trial with appropriately fit hearing aids worn on a full-time basis (8 hours per day)..
7. Patent cochlea and normal cochlear anatomy.
8. Must be in a habilitation/educational program with an emphasis on spoken language development.

Exclusion Criteria:

1.3 Criteria for Exclusion in Populations 1 and 2

1. Medical or psychological conditions that contraindicate undergoing surgery.
2. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
3. Unrealistic expectations on the part of the candidate and/or candidate's family, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices.
4. Unwillingness or inability of the candidate to comply with all investigational requirements.
5. Active middle ear infection.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2018-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Gantz, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult: Population 1: 15 Adults who have a severe sensorineural hearing loss with a pure-tone average (PTA) between 60-90 dB HL between 125-1500 Hz and profound loss at higher frequencies.
  Intervention: These patients will receive a Hybrid L24 cochlear implant.
  Cochlear® Nucleus™ Hybrid L24: The Nucleus Hybrid L24 cochlear implant incorporates an electrode array designed to preserve residual hearing. This has been accomplished by employing a thin, straight, intracochlear electrode array attached to a Nucleus cochlear implant receiver/stimulator. The Nucleus Hybrid L24 array has 22 electrodes spread over 16 mm and an anticipated insertion depth of 16 mm. It is slim, with its dimensions ranging from 0.35 x 0.25 mm (at the tip) to 0.55 x 0.4 mm, and designed to minimize lateral wall forces with a stiffened basal section to prevent buckling. The resultant insertion angle is about 280-300° in the scala tympani for the Hybrid L24, as confirmed in temporal bone trials at the Medical University Hannover and the University of Melbourne.
- Children and Adolescents (L24): Children (ages 5-12 years) and adolescents (ages 13-15 years) who have a sensorineural hearing loss with a pure-tone average (PTA) between 70-90 dB HL between 125-1500 Hz, a hearing threshold >90 dB HL at 1500 Hz and profound loss at higher frequencies.
  Intervention: These patients will receive a Hybrid L24 cochlear implant.
  Cochlear® Nucleus™ Hybrid L24: The Nucleus Hybrid L24 cochlear implant incorporates an electrode array designed to preserve residual hearing. This has been accomplished by employing a thin, straight, intracochlear electrode array attached to a Nucleus cochlear implant receiver/stimulator. The Nucleus Hybrid L24 array has 22 electrodes spread over 16 mm and an anticipated insertion depth of 16 mm. It is slim, with its dimensions ranging from 0.35 x 0.25 mm (at the tip) to 0.55 x 0.4 mm, and designed to minimize lateral wall forces with a stiffened basal section to prevent buckling. The resultant insertion angle is about 280-300° in the scala tympani for the Hybrid L24, as confirmed in temporal bone trials at the Medical University Hannover and the University of Melbourne.
- Children and Adolescents S12: Children (ages 5-12 years) and adolescents (ages 13-15 years) who have a sensorineural hearing loss with a pure-tone average (PTA) between 70-90 dB HL between 125-1500 Hz, a hearing threshold hearing threshold between 70-90 dB HL at 1500 Hz and profound loss at higher frequencies.
  Intervention: These patients will receive a Hybrid S12 cochlear implant.
  Cochlear® Nucleus™ Hybrid S12: The Nucleus Hybrid S12 cochlear implant incorporates an electrode array designed to stimulate the high-frequency, basal region of the cochlea while maintaining useful acoustic hearing in the low-frequency, apical region. This has been accomplished by employing a short, thin, straight intracochlear electrode array attached to a Nucleus cochlear implant receiver/stimulator. The electrode array incorporates a collar to prevent over-insertion, or further migration, into the cochlea beyond the point where the basal turn curves into the ascending segment. Thus, the electrode array is placed within the straight segment of the basal turn of the scala tympani via a cochleostomy.
Period: Overall Study
Arm/Group | Adult | Children and Adolescents (L24) | Children and Adolescents S12
Started | 15 | 5 | 0
Completed | 14 | 3 | 0
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: No children were enrolled and implanted with the S12 cochlear implant
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult | Children and Adolescents (L24) | Children and Adolescents S12 | Total
Number analyzed (Participants) | 15 | 5 | 0 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 5 |  | 5
  Between 18 and 65 years | 15 | 0 |  | 15
  >=65 years | 0 | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.7) | 13.04 (1.8) |  | 42.6 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 0 | 10
  Male | 9 | 1 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 00 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 15 | 5 | 0 | 20
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in CNC Word Perception
Description: Pre-operatively, speech perception testing will be conducted using the ear implanted and bilaterally with appropriately fit hearing aids. Post-operatively, speech perception testing will be attempted in the following conditions (unless otherwise noted):
  Combined stimulation (cochlear implant and any hearing aids worn on the implanted or non-implanted ears)
  Testing will be in quiet at 60 dB(A). The CNC word perception test consists of multiple lists of 50 3-syllable words (consonant-nucleus-consonant) that are presented through a loudspeaker using an open set format. Percent correct is calculated by the number of words identified by the subject out of the 50 words presented.
Time Frame: pre-op, 3, 6, 12, 24 months in the adults and pre-op, 3, 6, 12, 24, 36, 48, and 60 months post-implantation for children
Population: adults study testing was completed at 24 months
Measure: Mean (Standard Error); unit: percentage of words correct
Arm/Group | Adult | Children and Adolescents (L24) | Children and Adolescents S12
Number analyzed (Participants) | 15 | 5 | 0
percentage of words correct
  baseline (pre-op) | 27.6 (4.4) | 34 (5) |
  3 months | 55.9 (6.6) | 68 (7) |
  6 months: number analyzed (Participants) | 13 | 5 | 0
  6 months | 63.5 (6.4) | 64 (9) |
  12 months: number analyzed (Participants) | 13 | 5 | 0
  12 months | 66.7 (6.0) | 69 (7) |
  24 months: number analyzed (Participants) | 12 | 5 | 0
  24 months | 70.5 (7.5) | 67 (61) |
  36 months: number analyzed (Participants) | 0 | 4 | 0
  36 months |  | 61 (14) |
  48 months: number analyzed (Participants) | 0 | 3 | 0
  48 months |  | 62 (18) |
  60 months: number analyzed (Participants) | 0 | 3 | 0
  60 months |  | 65 (19) |

2. Secondary Outcome: Change in Localization
Description: Pre-operatively and post-operative, testing will be conducted using bilaterally fitted devices (preoperatively) and a cochlear implant and bilateral hearing aids (if applicable) postoperatively (combined condition). Everyday sounds will be presented from one of eight loudspeakers at 60 dBA forming a 108- arc. The participant will face the center of the speaker array at a 1.4 m. 16 different sounds will be repeated 6 times and presented randomly from one of the loudspeakers. Localization performance was calculated by the average root-mean-square (RMS) error in degrees.
Time Frame: Preoperatively and at 6 and 24 months post op in adults and pre op and 12 and 24 mos in children
Population: patient time and no children in the S12 study
Measure: Mean (Standard Error); unit: RMS Error in Degrees
Arm/Group | Adult | Children and Adolescents (L24) | Children and Adolescents S12
Number analyzed (Participants) | 15 | 4 | 0
RMS Error in Degrees
  preoperative (baseline): number analyzed (Participants) | 15 | 3 | 0
  preoperative (baseline) | 23 (2.1) | 18 (2.1) |
  6 months: number analyzed (Participants) | 13 | 4 | 0
  6 months | 34 (1.8) | 26 (3.8) |
  12 months: number analyzed (Participants) | 10 | 3 | 0
  12 months | 32 (2.5) | 24 (3.2) |

3. Secondary Outcome: AzBio +5 Noise
Description: Sentences in a +5 dB noise will be administered. Sentences will be tested at 60 dB(A) and noise at 55 dB(A) from the front. Pre-operatively, speech perception testing will be conducted using the ear implanted and bilaterally with appropriately fit hearing aids. Post-operatively, speech perception testing will be attempted in the following conditions (unless otherwise noted): Combined stimulation (cochlear implant and any hearing aids worn on the implanted or non-implanted ears) The AzBio sentence perception test consists of multiple lists of 20 sentences that are presented in sound-field from a loudspeaker using an open set format. Percent correct is calculated by the number of words correctly identified by the subject out of the total number of words presented in the sentence lists.
Time Frame: Adults pre-op, 3, 6, 12, 24 months post op
Population: protocol did not include testing on AzBio Sentences in noise with children/adolescents
Measure: Mean (Standard Error); unit: percentage of words in sentence
Arm/Group | Adult | Children and Adolescents (L24) | Children and Adolescents S12
Number analyzed (Participants) | 15 | 0 | 0
percentage of words in sentence
  preoperative (baseline) | 14.6 (5.04) |  |
  3 months: number analyzed (Participants) | 11 | 0 | 0
  3 months | 26.4 (4.9) |  |
  6 months: number analyzed (Participants) | 12 | 0 | 0
  6 months | 36.3 (6.7) |  |
  12 months: number analyzed (Participants) | 12 | 0 | 0
  12 months | 46.5 (5.6) |  |
  24 months: number analyzed (Participants) | 10 | 0 | 0
  24 months | 51.4 (7.8) |  |

ADVERSE EVENTS:
Time Frame: adults: preop through 24 months postop Children/adolescents: preop through 60 months postop
Description: same as clinicaltrials.gov
Arm/Group | Adult | Children and Adolescents (L24) | Children and Adolescents S12
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2011-09-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT01975571/Prot_000.pdf